CLINICAL TRIAL: NCT02151968
Title: Traditional Blind Versus Ultrasound-guided Peribulbar Blockade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Paul McHardy, Lecturer, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USG123
Record Dates: First submitted 2014-05-20; First posted 2014-06-02 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Retinal and Infra-ocular Pathology
MeSH Terms: interventions — Anesthesia, Local

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional blind peribulbar block (Active Comparator)
  Interventions: Procedure: Local Anaesthetic Injection
- Ultrasound-guided peribulbar block (Experimental)
  Interventions: Procedure: Local Anaesthetic Injection; Procedure: Ultrasound-Guidance

INTERVENTIONS:
Procedure: Local Anaesthetic Injection — Local anaesthetic is injected into the eye.
Procedure: Ultrasound-Guidance — Device: Ultrasound Machine
  Peribulbar block local anaesthetic is injected into the eye with ultrasound guidance.
  Other Names: Ultrasound Machine
  Arms: Ultrasound-guided peribulbar block

SUMMARY:
Eye surgeries are traditionally performed under local anaesthesia with a peribulbar block. This is a blind technique where local anaesthetic is injected into the back of the eye to make the eye numb and motionless for surgery. This is a blind injection and can be associated with complications such as bleeding, rupture of eye globe, blindness, increasing the pressure of the eye etc. It also has a high failure rate resulting in need for additional injections, further exposing the patient to possible complications. The investigators propose to perform the peribulbar block with ultrasound to guide the block needle placement and injection. The investigators hypothesize that ultrasound guided peribulbar blocks would have higher success rate (less need for additional injections) and that the total amount of local anaesthetics used would be decreased.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing vitrectomy surgery

Exclusion Criteria:

* Lack of informed consent
* Coagulopathic disorder, anticoagulated with INR (international normalized ratio) > 1.5 or platelet count less than 75 x 10^9/L
* Pathological myopia. Inability of patient to lie down for 2 hours for the operation -Local infection at site of needle entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Failure of peribulbar block | 10 minutes after block performed
  Ocular Anaesthetic Scoring System (OASS) score of less than 10 will be considered inadequate for surgery and a block failure.

SECONDARY OUTCOMES:
Quality of the block | 5 and 10 min after block performed
  Quality of the block based on the OASS score will be classified as poor (0-3), average (4-9) and good (10-14).
Incidence of Supplemental Peribulbar injections | Operative day 0
  To determine incidence of additional peribulbar injections after failure of original block as determined preoperatively by the anaesthetist or intraoperatively by the surgeon.
Volume of Total Local Anaesthetic Used | Operative day 0
  The total volume of local anaesthetic used for peribulbar block preoperatively and intraoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada